CLINICAL TRIAL: NCT03807765
Title: Phase Ib Study of Stereotactic Radiation and Nivolumab in the Management of Metastatic Breast Cancer Brain Metastases
Brief Title: Stereotactic Radiation and Nivolumab in the Management of Metastatic Breast Cancer Brain Metastases
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-19765; CA209-8NK (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2019-01-15; First posted 2019-01-17 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Breast Cancer; Brain Metastases
Keywords: breast cancer; brain metastases
MeSH Terms: conditions — Breast Neoplasms; Brain Neoplasms | interventions — Nivolumab; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Nivolumab followed by stereotactic radiosurgery (SRS) (Experimental): 480 mg Nivolumab will be given intravenously every 4 weeks, followed by SRS the week after the initial dose of Nivolumab.
  Interventions: Drug: Nivolumab; Radiation: Stereotactic Radiosurgery

INTERVENTIONS:
Drug: Nivolumab — 480 mg intravenous Nivolumab administered every 4 weeks.
  Other Names: Opdivo
Radiation: Stereotactic Radiosurgery — Patients will receive single session SRS to intact brain metastases and post-operative cavities.
  A linear accelerator (LINAC)-based frameless delivery system will be used to deliver the stereotactic radiation. The lesion will be defined using gadolinium enhanced MRI with 1 mm slices for treatment planning purposes prior to the delivery of radiation. The MRI image will be co-registered and fused with CT imaging. Doses will be prescribed to ensure coverage of at least 95% of the planning target volume (PTV) with the prescription dose. Treatments will be delivered using dynamic conformal arcs or intensity modulated radiotherapy.

SUMMARY:
This study is to find out if administration of stereotactic radiosurgery (SRS) given after Nivolumab will improve overall response rate/anti-tumor activity in patients with metastatic breast cancer with brain metastases.

ELIGIBILITY:
Inclusion Criteria:

* Provides signed and dated informed consent
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Age 18 or older
* Breast cancer with brain metastases, as documented by extracranial tumor biopsy with MRI brain imaging or intracranial surgical pathology revealing brain metastases
* 10 or less brain metastases eligible for SRS to brain metastases or to the post-operative bed
* Maximum diameter of the largest intact brain metastases ≤ 4 cm
* Eastern Cooperative Oncology Group performance status 0 to 2
* Prior treatment with taxane based chemotherapy with anthracyclines (if appropriate)
* A formalin-fixed, paraffin-embedded tumor tissue block or 10 unstained slides of intracranial/extracranial tumor sample (archival or recent) for biomarker evaluation should be made available and submitted to the central lab for correlative studies. If attempts to obtain archival tissue are unsuccessful the patient may be enrolled.
* Individuals with prior SRS/fractioned stereotactic radiotherapy (FSRT) treatment will be allowed if active measurable disease has not previously been treated with radiation therapy
* Continuing concurrent use of hormonal therapy or HER2-targeted therapy is allowed if the patient exhibits brain metastases progression during treatment
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin) within 24 hours prior to the administration of each dose of study agent.
* WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug(s), plus 5 half-lives of study drug (half-life up to 25 days), plus 30 days (duration of ovulatory cycle) for a total of 5 months after treatment completion.

Exclusion Criteria:

* Presence of leptomeningeal disease
* Prior whole brain radiation therapy
* All toxicities attributed to prior anticancer therapy must have been resolved to Grade 1 (NCI CTCAE Version 5) or baseline before administration of study drug(s) . Some exceptions apply.
* Women who are pregnant or breastfeeding
* Active, known, or suspected autoimmune disease. Patients with an autoimmune paraneoplastic syndrome requiring concurrent immunosuppressive treatment are excluded. Some exceptions apply.
* Prior therapy with antiPD-1, antiPD-L1, antiPD-L2, antiCD137, or antiCTLA-4 antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways)
* Interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity
* Any patient requiring supplemental oxygen therapy
* Patients with prior history of non-breast cancer malignancies are excluded except in the case of adequately treated basal cell cancer, squamous cell skin cancer, chronic lymphocytic leukemia, or other indolent diseases not requiring therapy
* Known medical condition that, in the investigator's opinion, would increase the risk associated with study participation or study drug(s) administration or that would interfere with the interpretation of safety results
* Major surgery or significant traumatic injury that has not been recovered from by 14 days before the initiation of study drug
* Current or prior participation in a study of an investigational agent or investigational device within 2 weeks of first dose of study treatment
* Positive test for: a. Hepatitis B virus using Hepatitis B virus surface antigen (Hepatitis B virus surface antigen) test b. Hepatitis C virus (HCV) using HCV ribonucleic acid or HCV antibody test that indicates acute or chronic infection c. Exception: Individuals with a positive test for HCV antibody but no detection of HCV ribonucleic acid indicating no current infection are eligible
* Medical history of testing positive for HIV or AIDS. No HIV testing is required, unless mandated by a local health authority.
* Inadequate hematologic function
* Inadequate hepatic function
* Inadequate pancreatic function
* History of allergy or hypersensitivity to any of the study drugs or study drug components
* Individuals who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2020-09-08 (Actual); Study Completion 2025-03-18 (Actual)

PRIMARY OUTCOMES:
Number of Participants who experience Dose Limiting Toxicities | Up to 8 weeks
  Neurologic dose limiting toxicities will be defined as: Symptomatic radionecrosis, >/= Grade 3 headache, >/= Grade 3 memory impairment, New onset >/= grade 3 seizures.
  3 participants will be enrolled with an 8 week safety observation period. If no patients develop unacceptable neurologic toxicity attributable to SRS, the study will proceed. If 1 patient develops unacceptable neurologic toxicity among the first 3, an additional 3 patients will be enrolled to determine the rate of unacceptable toxicity with 6 patients. If no more patients develop unacceptable neurologic toxicities among the first 6 patients, the study will proceed with a dose expansion of 6 patients.
  If 2 or more patients develop unacceptable neurologic toxicity among the first 3 or 6 patients, the dose of radiation therapy will be adjusted. If excessive toxicities are noted with radiation dose level -1, treatment will proceed with nivolumab alone.

SECONDARY OUTCOMES:
Evaluation of intracranial local brain tumor following treatment | At 3, 6 and 12 months post treatment
  Intracranial local brain tumor control following SRS and Nivolumab will be determined from irradiated lesions according to Response Assessment in Neuro-Oncology (RANO) criteria.
Evaluation of intracranial distant brain tumor following treatment | At 3, 6 and 12 months post treatment
  Intracranial distant brain tumor control following SRS and Nivolumab will be determined by the development of new lesions outside of the irradiated area.
Intracranial Progression Free Survival (PFS) | Up to 12 months
  Time from the date of start of treatment to the investigator-determined date of progression (determined by RANO) or death due to any cause, whichever occurs first.
Extracranial Progression Free Survival (PFS) | Up to 12 months
  Time from the date of start of treatment to the investigator determined date of progression (determined by Immune-Related Response Evaluation Criteria in Solid Tumors [irRECIST]) or death due to any cause, whichever occurs first.
Overall Survival | Up to 24 months
  Overall Survival defined as time from the date of start of treatment to death.

CONTACTS AND LOCATIONS:
Overall Officials: Kamran Ahmed, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ahmed KA, Kim Y, Kim S, Wang MH, DeJesus M, Arrington JA, Soyano AE, Armaghani AJ, Costa RLB, Loftus LS, Rosa M, Caudell JJ, Diaz R, Etame AB, Tran ND, Soliman H, Czerniecki BJ, Forsyth PA, Yu HM, Han HS. Nivolumab and stereotactic radiosurgery for patients with breast cancer brain metastases: long-term results and biomarker analysis from a non-randomized, open-label, phase Ib study. J Immunother Cancer. 2025 Apr 28;13(4):e011432. doi: 10.1136/jitc-2024-011432. PMID 40295143
- [Derived] Ahmed KA, Kim Y, Arrington JA, Kim S, DeJesus M, Soyano AE, Armaghani AJ, Costa RLB, Khong HT, Loftus LS, Rosa M, Caudell JJ, Diaz R, Robinson TJ, Etame AB, Tran ND, Sahebjam S, Soliman HH, Czerniecki BJ, Forsyth PA, Yu HM, Han HS. Nivolumab and Stereotactic Radiosurgery for Patients With Breast Cancer Brain Metastases: A Nonrandomized, Open-Label Phase 1b Study. Adv Radiat Oncol. 2021 Sep 11;6(6):100798. doi: 10.1016/j.adro.2021.100798. eCollection 2021 Nov-Dec. PMID 34934864
- See also: Moffitt Cancer Center Clinical Trials Website — https://moffitt.org/clinical-trials-research/clinical-trials/